CLINICAL TRIAL: NCT01587144
Title: An International, Multi-Center, Randomized, Double Blind Placebo Controlled Phase II Study to Evaluate the Safety and Efficacy of Lucanthone Administered as an Adjunct to Radiation and Temozolomide for Primary Therapy of Glioblastoma Multiforme
Brief Title: Safety and Efficacy Study of Lucanthone When Used in Combination With Temozolomide(TMZ) and Radiation to Treat Glioblastoma Multiforme(GBM)
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Sponsor's decision
Sponsor: Spectrum Pharmaceuticals, Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SPI-LUC-11-01
Record Dates: First submitted 2012-04-11; First posted 2012-04-30 (Estimated); Last update posted 2021-10-19 (Actual); Status verified 2021-10

CONDITIONS: Glioblastoma Multiforme
Keywords: GBM
MeSH Terms: conditions — Glioblastoma | interventions — Lucanthone; Temozolomide; Radiation

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Placebo (Placebo Comparator): Participants will receive a matching placebo as an adjunct in initial six weeks of concomitant therapy with TMZ and radiation, followed by a maintenance phase of six cycles of TMZ given on Days 1 to 5 of a 28-day cycle (+/- 3 days).
  Interventions: Drug: Temozolomide (TMZ); Radiation: Radiation; Drug: Placebo
- Lucanthone (Active Comparator): Participants will receive Lucanthone as an adjunct in initial six weeks of concomitant therapy with TMZ and radiation, followed by a maintenance phase of six cycles of TMZ given on Days 1 to 5 of a 28-day cycle (+/- 3 days).
  Interventions: Drug: Lucanthone; Drug: Temozolomide (TMZ); Radiation: Radiation

INTERVENTIONS:
Drug: Lucanthone — Lucanthone will be given as an oral at 10-15 mg/kg/day for 6 weeks during the concomitant phase. In the maintenance phase, placebo will be administered on days 1-5 of a 28-day cycle for 6 cycles.
  Arms: Lucanthone
Drug: Temozolomide (TMZ) — TMZ is administered at 75mg/m2 daily for 42 days during the concomitant phase. TMZ is administered for an additional 6 cycles of maintenance treatment. Dosage in Cycle 1 (maintenance) is 150 mg/m2 once daily for 5 days followed by 23 days without treatment.
  Cycles 2-6: At the start of Cycle 2, the dose can be escalated to 200 mg/m2, if the common terminology criteria (CTC) nonhematologic toxicity for Cycle 1 is Grade ≤2 (except for alopecia, nausea, and vomiting), absolute neutrophil count (ANC) is ≥1.5 x 109/L, and the platelet count is ≥100 x 109/L. The dose remains at 200 mg/m2 per day for the first 5 days of each subsequent cycle except if toxicity occurs.
Radiation: Radiation — 60 Gy administered in 30 fractions for 42 days in the concomitant phase.
Drug: Placebo — Placebo will be given as an oral at 10-15 mg/kg/day for 6 weeks during the concomitant phase. In the maintenance phase, placebo will be administered on days 1-5 of a 28-day cycle for 6 cycles.
  Arms: Placebo

SUMMARY:
The purpose of the study is to determine the effectiveness of an investigational drug called lucanthone, when combined with temozolomide (TMZ) and radiation in the treatment of Glioblastoma Multiforme (GBM).

DETAILED DESCRIPTION:
This is an international, multicenter, randomized, double blind placebo controlled phase II study to evaluate the safety and efficacy of lucanthone administered as an adjunct to patients receiving primary treatment of GBM with temozolomide and radiation. Eligible patients will be randomized to lucanthone or placebo arm in ratio of 1:1. The treatment period will be in two phases ; an initial six weeks of concomitant therapy with temozolomide and radiation, followed by a maintenance phase of six cycles of temozolomide given on Days 1 to 5 of a 28- day cycle (+/- 3 days). Lucanthone / placebo will be given as an add on in both concomitant and maintenance phases.

ELIGIBILITY:
Main Inclusion Criteria:

1. 18 and 70 years of age in India, 18 years and above in US
2. Histologically proven GBM who

   * May or may not have undergone surgery
   * Is scheduled to receive treatment with temozolomide and radiation.
3. Karnofsky score ≥ 70%.

Main Exclusion Criteria:

1. Diagnosis of recurrent brain tumor.
2. Received temozolomide previously.
3. Absolute neutrophil count ≤ 1.5 X 109/L.
4. Screening platelet count < 100 K/uL.
5. Screening bilirubin > 1.6 mg/dL.
6. Screening creatinine > 2.25 mg/dL in men and 1.8 mg/dL in women.
7. Screening ALT or AST > 2.5 times the upper limit of the laboratory reference range.
8. Unstable medical condition or significant comorbid pathophysiology (e.g. active infection, poorly controlled diabetes, unstable angina, severe heart failure) that would interfere with his/her participation in the study.
9. Enrolled, or plans to enroll, in a concurrent treatment protocol with another investigational product.
10. Receiving, or plans to receive, an anti-cancer therapy other than temozolomide during the study.
11. Received prior chemotherapy or radiation therapy within four weeks of enrollment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2012-06-19 (Actual); Primary Completion 2013-04-15 (Actual); Study Completion 2013-04-15 (Actual)

PRIMARY OUTCOMES:
Progression Free Survival | 9 months
  Progression Free Survival: defined as the time from randomization until objective tumor progression or death

SECONDARY OUTCOMES:
Objective response rate (ORR) | one year
  Fraction of patients with a Complete Response (CR) or Partial Response (PR) at anytime through the 12 months visit.
Overall Survival | one year
  Overall Survival: The time from randomization until death.
Safety Profile of Lucanthone | one year
  Safety Profile of Lucanthone at 10-15 mg/kg/day.

CONTACTS AND LOCATIONS:
Locations (10):
- United States (6):
  - UCSD Moores Cancer Center, La Jolla, California
  - UCI Medical Center, Orange, California
  - Dent Neurologic Institute, Amherst, New York
  - Fairview Hospital Moll Cancer Center/Cleveland Clinic, Cleveland, Ohio
  - Cleveland Clinic, Cleveland, Ohio
  - Hillcrest Hospital Hirsh Cancer Center/Cleveland Clinic, Mayfield, Ohio
- India (4):
  - Gujarat Cancer Research Institute, Ahmedabad, Gujarat
  - Jaslok Hospital & Research Centre, Mumbai, Maharashtra
  - Bhagwan Mahaveer Cancer Hospital & Reseach Centre, Jaipur, Rajasthan
  - Chittaranjan National Cancer Institute, Kolkata, West Bengal